CLINICAL TRIAL: NCT03656926
Title: A Phase III Clinical Trial to Demonstrate Efficacy / Safety of Liposomal Cyclosporine A + Standard of Care (SoC) vs SoC Alone in Treating Chronic Lung Allograft Dysfunction / Bronchiolitis Obliterans in Patients Post Double Lung Transplant
Brief Title: Efficacy + Safety of Liposome Cyclosporine A to Treat Bronchiolitis Obliterans Post Double Lung Transplant (BOSTON-2)
Acronym: BOSTON-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT - L-CsA - 302 - DLT; 2018-003205-25 (EudraCT Number)
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Bronchiolitis Obliterans; Chronic Rejection of Lung Transplant; Lung Transplant Rejection; Lung Transplant; Complications; Lung Transplant Failure and Rejection; Chronic Lung Allograft Dysfunction
MeSH Terms: conditions — Bronchiolitis Obliterans; Rejection, Psychology | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-CsA treatment plus SoC (Experimental): Liposomal Cyclosporine A (L-CsA) 10 mg twice daily for 48 weeks, plus Standard of Care Therapy
  Interventions: Drug: Liposomal Cyclosporine A
- Standard of Care (Active Comparator): This is a maintenance regimen of immunosuppressive agents
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Liposomal Cyclosporine A — This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm.
  The L-CsA was administered as 10 mg/2.4 mL inhalation via the PARI eFlow device BID (morning/evening, approximately 12 hours apart) for 48 weeks. Nebulization time per inhalation dose was approximately 6 to 17 minutes.
  Patients received training on the use of the device and the first dose of L-CsA was self-administered by each patient under the supervision of trained personnel. In addition, during all subsequent scheduled visits the L-CsA inhalation was self-administered by the patient and under the supervision of trained study personnel.
  Other Names: L-CsA
  Arms: L-CsA treatment plus SoC
Drug: Standard of Care — Standard of Care Therapy (SoC). The SoC included maintenance immunosuppressive medication including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent; but also a prophylaxis against common opportunistic infections, and all other necessary medications and therapies for the optimal care of the patient.
  This also included vaccination against COVID-19 All changes in concurrent treatment or medication were administered according to site's SoC.
  The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, should be on a stable regimen for a least 4-weeks prior to randomization and continued to receive azithromycin during the trial as deemed appropriate by the investigator.
  Other Names: SoC
  Arms: Standard of Care

SUMMARY:
The objective of this trial was to assess the efficacy and safety of aerosolized liposomal cyclosporine A (L-CsA) as add-on therapy to standard of care (SoC) as compared to SoC alone in double lung transplant (DLT) recipients with chronic lung allograft dysfunction (CLAD)-bronchiolitis obliterans syndrome (BOS).

DETAILED DESCRIPTION:
This was a Phase III, open-label, prospective, multicenter, randomized, controlled clinical trial of L-CsA for the treatment of BOS in adults following DLT. The patient population was recipients of a double pulmonary allograft, > or = 18 years old, with clinically defined CLAD--BOS with screening FEV1 >or = 51% of personal best FEV1 value post-transplant during the Screening period.

The rationale for an open-label study was driven by concerns that a sucrose-containing placebo formulation could increase a potential risk of pulmonary infection without the benefit of L-CsA. Sucrose is a lyoprotectant in the manufacturing process. After carefully considering alternative options for lyoprotection, no sugar-free alternatives that would qualify as a real placebo (i.e., undistinguishable by means of appearance, taste, or smell) could be identified.

Therefore, an open-label, randomized controlled trial versus SoC was the only suitable alternative.

An open-label clinical trial generally bears the potential for bias in patient treatment and care, and thus trial outcome. However, for this trial the risk of bias is considered low because of the following reasons:

* During the trial, the general treatment of BOS was use of immunosuppressive therapy to the highest tolerable level unless limited by systemic toxicity. As inhaled L-CsA has not been associated with additional systemic drug burden, dose reductions or adaptations of other components of the immunosuppressive cocktail would not be required and were not desired.
* The selected primary endpoint FEV1 is an objective parameter and its measurement was performed according to recommended guidelines of American Thoracic Society (ATS)/European Respiratory Society (ERS) which had to be respected by each participating center. Following this methodology, a subjective and intentional manipulation of outcome was highly unlikely even if healthcare professional and patient were aware of the treatment allocation.
* Pulmonary function technicians, respiratory therapists, or physiotherapists who performed spirometry at each site were blinded to each patient's study treatment assignment.
* Finally, the correctness and validity of individual FEV1 curves and their resulting value had to be approved in a central and blinded reading by a pulmonary expert who was independent and not involved in patient care or treatment. The implementation of these measures should have ensured that the reported data of the primary outcome was as free as possible of bias induced by the open-label trial design.

Stratification prior to randomization was performed to limit imbalances between treatment arms with respect to key variables and potential confounders.

There were major recruitment issues in both the BOSTON-1 trial (SLT recipients) and the present BOSTON-2 trial, in part due to Coronavirus disease-2019 (COVID-19) and specifically in BOSTON-1 due to a marked decline over time in the use of SLT. Following FDA recommendation to obtain an adequately sized safety database for inhaled L-CsA and reach the originally planned sample size for BOSTON-1 and BOSTON-2 trials combined, it was planned to stop randomization into the two Phase III clinical trials upon achievement of a combined total of approximately 220 patients, of which approximately 160 to 170 patients were planned for enrollment in BOSTON-2. To assure balance between treatment arms with regard to key variables and potential confounders, stratification prior to randomization was performed. Within each of the 8 strata, using a permuted blocks randomization, patients were randomly assigned with equal probability (1:1) to receive either L-CsA (10 mg) via the PARI eFlow Nebulizer System twice daily (BID) plus SoC treatment or SoC alone, for a period of 48 weeks. Patients were monitored every 4 to 8 weeks over 48 weeks for efficacy parameters and for all safety evaluations. All patients were eligible to continue in an open-label extension trial of L-CsA, BOSTON-3 (Study BT-L-CsA-303-FU) following completion of either BOSTON-1 or BOSTON-2.

Up to 11 visits (Screening, V1 through V10) were planned during the clinical trial. After informed consent had been obtained, a Screening Visit was carried out to check general eligibility for participation. At the Baseline Visit (V1, Randomization Visit), inclusion and exclusion criteria were re-checked, and Baseline serial spirometry was performed. During the 48-week treatment period, visits were scheduled every 4 to 8 weeks (V2 to V9). Visit 9 (End of Treatment [EoT) was scheduled to occur 48 weeks after Visit 1. If a patient had an event that met the first criterion for progression of BOS, progression of BOS must have been confirmed by measurements that were taken with COMPACT spirometer at least 2 weeks apart. Visit 10 (EoS) was a safety follow-up visit performed 4 weeks after Visit 9/EoT only in patients not rolling over to the extension study (BOSTON-3). For patients who rolled over to BOSTON-3, the EoT Visit was the EoS Visit. Every effort was made to have all planned and unscheduled visits at the study site. However, if one of the visits from Visit 2 to Visit 8 and discontinuation visits could not be performed at the site due to COVID-19, remote visits (e.g., by telephone) were possible. Mandatory on-site visits were Screening Visit, Visit 1, and Visit 9.

ELIGIBILITY:
Inclusion Criteria:

Patients who met the following criteria as stated in the protocol were included in the study:

1. Adult patients of > or = 18 years who received a DLT at least 12 months prior to Screening.
2. Patients with BOS diagnosis defined as CLAD-BOS phenotype with:

   1. screening FEV1 between 51% and 85% of personal best FEV1 value post-transplant OR
   2. screening FEV1 > 85% of personal best FEV1 associated with EITHER a > or = 200 mL decrease in FEV1 in the previous 12 months OR according to medical history showing BOS progression.
3. Diagnosis of CLAD-BOS must have been made at least 12 months after lung transplantation and

   1. within 12 months prior to the Screening Visit OR
   2. more than 12 months from Screening and patient must have shown a decline in FEV1 >or = 200 ml in the previous 12 months before Screening, which was not due to acute infection or acute organ rejection.
4. Patients in whom the diagnosis of BOS had been confirmed by the elimination of other possible causes of obstructive or restrictive lung disease CLAD - restrictive allograft syndrome (RAS) phenotype.
5. Patients should have been on a drug maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must have been stable within 4 weeks prior to randomization with respect to the therapeutic agents. In case a patient was also receiving concomitant azithromycin for prophylaxis or treatment of BOS, in addition to the previously described immunosuppressive regimen, azithromycin must have been on a stable regimen for at least 4 weeks prior to randomization.
6. Patients capable of understanding the purposes and risks of the clinical trial, who had given written informed consent and agreed to comply with the clinical trial requirements/visit schedules, and who were capable of aerosol inhalation. Patients must have consented to retrieve prespecified data from the historic medical record (e.g., information related to the transplant surgery; spirometry data; medication use).
7. Women of childbearing potential must have had a negative serum or urine pregnancy test within 7 days prior to randomization and must have agreed to use one of the methods of contraception listed in Appendix II of the protocol in Appendix 16.1.1 through their EoS Visit.
8. Patients had no concomitant diagnoses that were considered fatal within one year (12 months) of Screening.

Exclusion Criteria:

1. Patients with confirmed other causes for loss of lung function, such as acute infection, acute rejection, restrictive allograft syndrome (RAS) (CLAD - RAS phenotype, see Protocol Specific Definition ), etc.
2. Cystic Fibrosis patients with multi-drug resistant infections not responding to available anti-microbial therapies.
3. Patients with acute antibody-mediated rejection at Screening. In this context, clinically stable patients (as judged by the Investigator) with detectable levels of donor specific antibodies (DSA) at the Screening Visit are eligible for the study.
4. Active acute bacterial, viral, or fungal infection not successfully resolved at least 4 weeks prior to the Screening Visit. Patients with chronic infection or colonization who are clinically stable as per judgement of the Investigator are eligible for the study.
5. Mechanical ventilation (including CPAP) within 12 weeks prior to Randomization.
6. Patients with uncontrolled hypertension.
7. Patient has baseline resting oxygen saturation of < 89% on room air or use of supplemental oxygen at rest.
8. Evidence of functional airway stenosis (e.g., bronchomalacia/tracheomalacia, airway stents, or airways requiring balloon dilatations to maintain patency) with onset after the initial diagnosis of BOS and ongoing at Screening and/or Randomization Visit.
9. Known hypersensitivity to L-CsA or to cyclosporine A.
10. Patients with chronic renal failure, defined as serum creatinine > 2.5 mg/dL at screening, or requiring chronic dialysis.
11. Patients with liver disease and serum bilirubin > 3-fold upper limit of normal range or transaminases > 2.5 upper limit of normal range.
12. Patients with active malignancy within the previous 2 years, including post-transplant lymphoproliferative disorder, with the exception of treated, localized basal and squamous cell carcinomas.
13. Pregnant women or women who are unwilling to use appropriate birth control to avoid pregnancy through their End of Study Visit.
14. Women who are currently breastfeeding.
15. Receipt of an investigational drug as part of a clinical trial within 4 weeks prior to the Screening Visit. This is defined as any treatment that is implemented under an Investigational New Drug (IND) or compassionate use.
16. Patients who have received extracorporeal photophoresis (ECP) for treatment of BOS within 1 month prior to Randomization.
17. Patients who are currently participating in an interventional clinical trial.
18. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures.
19. Any co-existing medical condition that in the Investigator's judgment will substantially increase the risk associated with the patient's participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Castellani, MD, Study Director — Zambon SpA, Chief Medical Officer and R&D
Locations (40):
- United States (21):
  - Banner Health, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Stanford University Hospital, Palo Alto, California
  - UC San Francisco, San Francisco, California
  - University of Florida Medical Center, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - CHU Erasme, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
- Copenhagen University Hospital, Copenhagen, Denmark
- France (3):
  - Marie-Lannelongue, Le Plessis-Robinson
  - CHU Hopital Nord, Marseille
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (2):
  - Hannover Medical School, Hanover
  - LMU Klinikum Großhadern, Munich
- Rabin Medical Center, Petah Tikva, Israel
- Spain (7):
  - Complexo Hospitalario de A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Marques de Valdecilla, Santander
  - University Hospital LA Fe, Valencia
- United Kingdom (2):
  - Royal Papworth Hospital, Cambridge
  - University of Manchester, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The COVID-19 pandemic impacted the conduct of the study. Based on the evolution of the outbreak and in accordance with country- and site-specific determinations, recruitment was put on hold starting on 20 March 2020.
  Recruitment was subsequently resumed in Quarter 3 2020. COVID- 19 might have affected the results for different reasons including changes in infection rate and type, quarantining, social distancing, and other considerations linked to different ways each site managed the pandemic.
Groups:
- L-CsA Treatment Plus SoC: Liposomal Cyclosporine A (L-CsA) 10 mg twice daily for 48 weeks, plus Standard of Care Therapy
  Liposomal Cyclosporine A: This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm.
  The L-CsA was administered as 10 mg/2.4 mL inhalation via the PARI eFlow device BID (morning/evening, approximately 12 hours apart) for 48 weeks. Nebulization time per inhalation dose was approximately 6 to 17 minutes.
  Patients received training on the use of the device and the first dose of L-CsA was self-administered by each patient under the supervision of trained personnel. In addition, during all subsequent scheduled visits the L-CsA inhalation was self-administered by the patient and under the supervision of trained study personnel.
- Standard of Care: This is a maintenance regimen of immunosuppressive agents
  Standard of Care: Standard of Care Therapy (SoC). The SoC included maintenance immunosuppressive medication including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent; but also a prophylaxis against common opportunistic infections, and all other necessary medications and therapies for the optimal care of the patient.
  This also included vaccination against COVID-19 All changes in concurrent treatment or medication were administered according to site's SoC.
  The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, should be on a stable regimen for a least 4-weeks prior to randomization and continued to receive azithromycin during the trial as deemed appropriate by the investigator.
Period: Overall Study
Arm/Group | L-CsA Treatment Plus SoC | Standard of Care
Started | 84 | 85
Full analysis set | 84 | 85
Safety analysis set | 84 | 85
Per protocol set | 46 | 70
Completed | 69 | 79
Not Completed | 15 | 6
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Screen fail after randomization | 1 | 0
Not completed — PI decision due to patient condition | 1 | 0
Not completed — Patient unresponsiveness | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS was defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized. All primary, secondary and exploratory endpoints were performed using the FAS, unless otherwise specified.
Groups:
- L-CsA Treatment Plus SoC - SAF: Liposomal Cyclosporine A (L-CsA) 10 mg twice daily for 48 weeks, plus Standard of Care Therapy
  Liposomal Cyclosporine A: This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm.
  The L-CsA was administered as 10 mg/2.4 mL inhalation via the PARI eFlow device BID (morning/evening, approximately 12 hours apart) for 48 weeks. Nebulization time per inhalation dose was approximately 6 to 17 minutes.
  Patients received training on the use of the device and the first dose of L-CsA was self-administered by each patient under the supervision of trained personnel. In addition, during all subsequent scheduled visits the L-CsA inhalation was self-administered by the patient and under the supervision of trained study personnel.
- Standard of Care - SAF: This is a maintenance regimen of immunosuppressive agents
  Standard of Care: Standard of Care Therapy (SoC). The SoC included maintenance immunosuppressive medication including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent; but also a prophylaxis against common opportunistic infections, and all other necessary medications and therapies for the optimal care of the patient.
  This also included vaccination against COVID-19 All changes in concurrent treatment or medication were administered according to site's SoC.
  The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, should be on a stable regimen for a least 4-weeks prior to randomization and continued to receive azithromycin during the trial as deemed appropriate by the investigator.
- Total: Total of all reporting groups
Arm/Group | L-CsA Treatment Plus SoC - SAF | Standard of Care - SAF | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 64 | 122
  >=65 years | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.69) | 56.2 (10.82) | 56.3 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 42 | 76
  Male | 50 | 43 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 75 | 70 | 145
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 2 | 8 | 10
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 3 | 5
  Belgium | 4 | 2 | 6
  United States | 30 | 31 | 61
  Denmark | 1 | 3 | 4
  United Kingdom | 3 | 3 | 6
  Israel | 4 | 1 | 5
  France | 4 | 8 | 12
  Germany | 15 | 19 | 34
  Spain | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in FEV1 (Liters) From Baseline to Week 48
Description: FEV1 is the Forced Expiratory Volume in One Second. The FEV1 data collected from the on-site COMPACTTM spirometer were to be considered primary, while data collected with the In2itiveTM home spirometer were to be used for supportive analyses.
Time Frame: Week 48
Population: Full analysis set: The FAS was defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized. Please note that N = number of patients in analysis set (N=84 for L-CSA + SoC and N=85 for SoC alone); n = number of patients with data available (n=64 for L-CSA + SoC and n=80 for SoC alone)
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- L-CsA Treatment Plus SoC - FAS: Liposomal Cyclosporine A (L-CsA) 10 mg twice daily for 48 weeks, plus Standard of Care Therapy
  Liposomal Cyclosporine A: This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm.
  The L-CsA was administered as 10 mg/2.4 mL inhalation via the PARI eFlow device BID (morning/evening, approximately 12 hours apart) for 48 weeks. Nebulization time per inhalation dose was approximately 6 to 17 minutes.
  Patients received training on the use of the device and the first dose of L-CsA was self-administered by each patient under the supervision of trained personnel. In addition, during all subsequent scheduled visits the L-CsA inhalation was self-administered by the patient and under the supervision of trained study personnel.
- Standard of Care - FAS: This is a maintenance regimen of immunosuppressive agents
  Standard of Care: Standard of Care Therapy (SoC). The SoC included maintenance immunosuppressive medication including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent; but also a prophylaxis against common opportunistic infections, and all other necessary medications and therapies for the optimal care of the patient.
  This also included vaccination against COVID-19 All changes in concurrent treatment or medication were administered according to site's SoC.
  The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, should be on a stable regimen for a least 4-weeks prior to randomization and continued to receive azithromycin during the trial as deemed appropriate by the investigator.
Arm/Group | L-CsA Treatment Plus SoC - FAS | Standard of Care - FAS
Number analyzed (Participants) | 64 | 80
Liters | -0.096 (0.1120) | -0.067 (0.1147)
Statistical Analysis 1: Comparison: L-CsA Treatment Plus SoC - FAS vs Standard of Care - FAS; V9 - week 48; Test type: Superiority — Estimates are from a Linear Mixed Model on the response variable change from baseline in FEV1 with factors for time splines, treatment, the interactions of time splines by treatment, baseline FEV1, the interactions of time splines with baseline FEV1, region (North America vs all other countries together), age (<55 versus >=55 years), use of azithromycin at randomization, and time as random effect; p = 0.6639, Mixed Models Analysis — This is a 1-side p value; least square mean difference = -0.028, 95% CI 2-sided [-0.160 to 0.104]

2. Secondary Outcome: Mean Change in FEV1/ Forced Vital Capacity (FVC) From Baseline to Week 48
Description: Forced Expiratory Volume in One Second on Forced Vital Capacity. It was analysed in the FAS using a LMM for repeated measurements, with baseline FEV1/FVC among covariates. In case of death or re- transplantation events, FEV1/FVC was imputed as zero at each nominal day post event. FEV1/FVC is a calculated ratio used to diagnose obstructive and restrictive lung disease. It represents the proportion of a patient's vital capacity that he/she is able to expire in the first second of forced expiration to the full forced vital capacity.
Time Frame: Week 48
Population: The FAS is defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized. All primary and secondary endpoints were performed using the FAS, unless otherwise specified. The number of patients with data available (n) for this outcome was 64 for L-Csa + SoC and 80 for SoC alone, while the number of patients (N) in the FAS is 84 and 85 respectively.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | L-CsA Treatment Plus SoC - FAS | Standard of Care - FAS
Number analyzed (Participants) | 64 | 80
ratio | -0.100 (0.0722) | -0.083 (0.0702)
Statistical Analysis 1: Comparison: L-CsA Treatment Plus SoC - FAS vs Standard of Care - FAS; Estimates were from a Linear Mixed Model on the response variable change from baseline in FEV1/FVC with factors for time splines, treatment, the interactions of time splines by treatment, baseline FEV1/FVC, the interactions of time splines with baseline FEV1/FVC, region (North America versus all other countries together), age (<55 versus > or = 55), use of azithromycin at randomization, and time as random effect; Test type: Superiority; p = 0.7792, Mixed Models Analysis; least square mean difference = -0.016, 95% CI 2-sided [-0.057 to 0.025]

3. Secondary Outcome: Time to Progression of Bronchiolitis Obliterans Syndrome (BOS)
Description: Time to progression of BOS, defined as the earliest of the following:
  * Absolute decrease from Baseline in FEV1 ≥10% or ≥ 200 mL (0.2 L) and absolute decrease in FEV1/FVC of > 5% OR
  * Worsening of BOS grade, OR
  * Re-transplantation, OR
  * Death from respiratory failure. More than one type of event might correspond to the event of BOS progression (even those occurring on the same date). In case progression of BOS was defined by more than one criterion on different dates, the earliest event date was considered, i.e., the date closer to randomization was used as the progression date.
Time Frame: From date of randomization until the date of first documented progression of BOS, or date of retransplantation, or date of death from respiratory failure, whichever came first, assessed up to 48 weeks.
Population: Full analysis set: The FAS was defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | L-CsA Treatment Plus SoC - FAS | Standard of Care - FAS
Number analyzed (Participants) | 84 | 85
weeks | NA [NA to NA] — Median and confidence interval limits were not achieved due to the low number of events | NA [NA to NA] — Median and confidence interval limits were not achieved due to the low number of events
Statistical Analysis 1: Comparison: L-CsA Treatment Plus SoC - FAS vs Standard of Care - FAS; For the statistical analysis, the estimand was the log hazard ratio of the L-CsA + SoC group relative to the SoC alone group. The treatment policy strategy was adopted for handling the IEs of treatment discontinuation. Dropouts due to other reasons and death from respiratory failure were to be treated as non-informative censoring; Test type: Superiority; p = 0.3110, Regression, Cox — 1-sided p value. The adjusted hazard ratio was calculated using Cox proportional hazards model, with covariates of treatment, age (< 55 vs > or= 55 years) with Efron's method of tie handling; adjusted hazard ratio = 1.19, 95% CI 2-sided [0.589 to 2.420]

4. Other Pre Specified Outcome: Acute Tolerability of L-CsA: FEV1 Change From Pre-dose to 1 Hour and 4 Hours Post-dose
Description: Acute tolerability of IMP (L-CsA) during initial dosing was determined by measuring spirometry 1 hour and 4 hours after treatment. The FEV1 was measured prior to dosing with L-CsA. A decline of ≥20% associated with symptoms could have warranted IMP discontinuation. Parameters reflecting acute tolerability of IMP were: spirometry, cough, or dyspnea.
Time Frame: Pre-dose and 1- and 4-hours post-dose on Visit 1
Population: SAF: The SAF was defined as all randomized patients receiving SoC and/or at least one dose of L-CsA, independently of the treatment allocation at randomization. All safety and tolerability data were summarized and analyzed using the SAF. Please note that only 77 patients had available data at 1 hour after treatment and only 72 had data 4h after treatment.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | L-CsA Treatment Plus SoC - SAF
Number analyzed (Participants) | 84
Liters
  1h post-dose | -0.019 (0.0855)
  4h post-dose | -0.005 (0.0914)

5. Other Pre Specified Outcome: Count of Participants With at Least One Adverse Event (AE)
Description: An untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine.
Time Frame: Baseline through study completion (52 weeks)
Population: SAF: The SAF was defined as all randomized patients receiving SoC and/or at least one dose of L-CsA, independently of the treatment allocation at randomization.
  Independently of the treatment allocation at randomization, patients were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care SAF: This is a maintenance regimen of immunosuppressive agents
  Standard of Care: Standard of Care Therapy (SoC). The SoC included maintenance immunosuppressive medication including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent; but also a prophylaxis against common opportunistic infections, and all other necessary medications and therapies for the optimal care of the patient.
  This also included vaccination against COVID-19 All changes in concurrent treatment or medication were administered according to site's SoC.
  The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, should be on a stable regimen for a least 4-weeks prior to randomization and continued to receive azithromycin during the trial as deemed appropriate by the investigator.
Arm/Group | L-CsA Treatment Plus SoC - SAF | Standard of Care SAF
Number analyzed (Participants) | 84 | 85
Participants
  with any TEAE | 73 | 77
  with any TEAE Leading to discontinuation of study treatment | 12 | 0
  with any TEAE Leading to study discontinuation | 5 | 3
  with any TEAE Leading to death | 2 | 4
  with any TEAE mild | 66 | 68
  with any TEAE moderate | 50 | 56
  with any TEAE severe | 21 | 18
  with any study treatment-related TEAE | 39 | 0
  with any serious TEAE | 46 | 44

ADVERSE EVENTS:
Time Frame: From baseline throughout the study, till week 52.
Description: Serious TEAEs by System Organ Class and Preferred Term in Safety Analysis Set are Reported by at Least 2 Patients Overall. Non serious adverse events are reported with a 0% threshold on the same set.
Arm/Group | L-CsA Treatment Plus SoC - SAF | Standard of Care - SAF
All-Cause Mortality (participants affected / at risk) | 2/84 | 4/85
Serious Adverse Events (participants affected / at risk) | 46/84 | 44/85
Other Adverse Events (participants affected / at risk) | 73/84 | 77/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA Treatment Plus SoC - SAF (N=84) | Standard of Care - SAF (N=85)
COVID-19 (Infections and infestations) | 23 (23) | 21 (23)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (6)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 0 (0) | 2 (2)
Transplant rejection (Immune system disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA Treatment Plus SoC - SAF (N=84) | Standard of Care - SAF (N=85)
COVID-19 (Infections and infestations) | 23 (23) | 21 (23)
Bronchitis (Infections and infestations) | 8 (9) | 5 (6)
Nasopharyngitis (Infections and infestations) | 6 (7) | 8 (9)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (4) | 4 (5)
Herpes Zoster (Infections and infestations) | 3 (3) | 4 (4)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral infection (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 3 (4)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pustule (Infections and infestations) | 1 (2) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 4 (5)
Superinfection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Bordetella infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Genital Herpes (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 7 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (6)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Throat clearing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 16 (18) | 15 (20)
Oedema peripheral (General disorders) | 7 (8) | 7 (7)
Fatigue (General disorders) | 5 (5) | 2 (2)
Pyrexia (General disorders) | 4 (7) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Barret's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukoplakia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyposmia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy perypheral (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 4 (4)
Renal impairment (Renal and urinary disorders) | 4 (4) | 1 (1)
Chronic kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (4)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 3 (3) | 2 (2)
Actinomyces test positive (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Drug level increased (Investigations) | 1 (1) | 0 (0)
Eosinophil count decreased (Investigations) | 1 (1) | 0 (0)
Forced expiratory volume abnormal (Investigations) | 1 (1) | 0 (0)
Fungal test positive (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haptoglobin increased (Investigations) | 1 (2) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Monocyte count increased (Investigations) | 1 (2) | 0 (0)
Neutrophil count increased (Investigations) | 1 (2) | 0 (0)
White blood cell count increased (Investigations) | 1 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Bronchoscopy (Investigations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Vitamin D increased (Investigations) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (4)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 2 (2) | 3 (3)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Sleeep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alpha-1 antitrypsin deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT03656926/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT03656926/SAP_001.pdf